CLINICAL TRIAL: NCT02449681
Title: A Phase 2 Study of Tarloxotinib (TH-4000) in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck or Skin
Brief Title: Study for Treatment of Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck or Skin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Rain Oncology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-602
Record Dates: First submitted 2015-05-12; First posted 2015-05-20 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Head-and-neck Squamous-cell Carcinoma
Keywords: squamous cell carcinoma; the head and neck; skin; TH-4000; Hypoxia; Tarloxotinib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Hypoxia

STUDY DESIGN:
Intervention Model Description: Open-label single arm two-stage, phase-2 study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TH-4000 (Tarloxotinib) (Experimental): TH-4000 150 mg/m2 will be administered by IV infusion over 60 minutes on Days 1, 8, 15 and 22 of each 28-day cycle until progressive disease (PD) or unacceptable toxicity.
  Interventions: Drug: TH-4000 (Tarloxotinib)

INTERVENTIONS:
Drug: TH-4000 (Tarloxotinib)
  Other Names: Tarloxotinib

SUMMARY:
This phase 2 study is designed to evaluate the safety and activity of TH-4000, a hypoxia-activated prodrug in participants with recurrent or metastatic squamous cell carcinoma of the head and neck or skin.

DETAILED DESCRIPTION:
An open label, multi-center Phase 2 study in which the pharmacokinetics, safety, tolerability and efficacy of TH-4000 will be assessed in participants with recurrent or metastatic squamous cell carcinoma of the head and neck or skin.

Hypoxia PET scans will be obtained in select centers to analyze potential predictors of tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Confirmed squamous cell carcinoma (SCC) of the head and neck (oropharynx, oral cavity, hypopharynx, or larynx) or skin
* For patients with oropharyngeal cancer, p16 status is known or can be determined
* Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Acceptable laboratory results as indicated by protocol
* Acceptable cardiac function as indicated by protocol

Exclusion Criteria:

* Received prior epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI) therapy for recurrent or metastatic Squamous Cell Carcinoma (e.g., oral EGFR TKIs such as erlotinib, gefitinib, or afatinib)
* Family history of long corrected QT interval (QTc) syndrome
* Receiving medication that prolongs QT interval ,with a risk of causing Torsades de Pointes (TdP), unless ECG meets inclusion criteria while on a stable dose of the medication
* Family history of long QTc syndrome
* Symptomatic central nervous system (CNS) lesions, or CNS lesions that require therapy
* Radiation therapy within 2 weeks prior to the first dose of study medication
* Major surgery within 4 weeks or minor surgery within 2 weeks prior to the first dose of study medication
* Concurrent active malignancy requiring systemic treatment
* Any other serious uncontrolled medical disorders or psychological conditions that may interfere with study conduct including but not limited to: clinically significant active infection
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with response rate as evaluated by RECIST criteria | Approximately 12 months

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose
Type of adverse events (AEs) | Up to 30 days after last dose
Severity of adverse events (AEs) | Up to 30 days after last dose
Duration of response (DOR) calculated for all patients achieving an objective response | Approximately 12 months
Progression-free survival (PFS) | Approximately 12 months
Overall Survival (OS) | Approximately 12 months
Maximum plasma concentration of TH-4000 (prodrug) and TH-4000E (TKI effector) | Cycle 1 Day 1 predose and up to 24 hours postdose
Area under the plasma concentration versus time curve of TH4000 (prodrug) and TH-4000E (TKI effector) | Cycle 1 Day 1 predose and up to 24 hours postdose
QTc Interval | Screening, Cycle 1 Day 1, 8, 15 & 22, Day 1 and study Termination

OTHER OUTCOMES:
Hypoxic volume as measured by Positron Emission Tomography (PET) hypoxia imaging | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Liu, Principal Investigator — Georgetown University Hospital Cancer Center
Locations (10):
- United States (8):
  - University of Southern California-Norris, Los Angeles, California
  - Stanford school of Medicine, Stanford, California
  - Georgetown Medical Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Walter Reed National Military Cancer Center, Bethesda, Maryland
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center (VICC), Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Peter MacCallum, East Melbourne, Victoria

REFERENCES:
- [Derived] McLean LS, Morris TA, Gramza A, Liu S, Khan SA, Colevas AD, Pearce T, Rischin D. A phase II study of tarloxotinib (a hypoxia activated prodrug of a pan-erb tyrosine kinase inhibitor) in patients with recurrent or metastatic squamous cell carcinoma of the head and neck or skin. Invest New Drugs. 2022 Aug;40(4):782-788. doi: 10.1007/s10637-022-01230-w. Epub 2022 Apr 18. PMID 35435625